CLINICAL TRIAL: NCT03725722
Title: A Phase 2b, Double-blind, Randomised, 5-arm, Vehicle-controlled, Dose Ranging Trial to Evaluate the Efficacy and Safety of Twice Daily Topical Applications of Delgocitinib Cream 1, 3, 8, 20 mg/g for 8 Weeks in Adult Subjects With Mild to Severe Atopic Dermatitis.
Brief Title: Dose-ranging Trial to Evaluate Delgocitinib Cream 1, 3, 8, and 20 mg/g Compared to Delgocitinib Cream Vehicle Over an 8-week Treatment Period in Adult Subjects With Atopic Dermatitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0133-1275
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Delgocitinib cream 1 mg/g (Experimental): Delgocitinib cream applied twice daily for 8 weeks
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 3 mg/g (Experimental): Delgocitinib cream applied twice daily for 8 weeks
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 8 mg/g (Experimental): Delgocitinib cream applied twice daily for 8 weeks
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream 20 mg/g (Experimental): Delgocitinib cream applied twice daily for 8 weeks
  Interventions: Drug: Delgocitinib cream
- Delgocitinib cream vehicle (Placebo Comparator): Delgocitinib cream vehicle applied twice daily for 8 weeks
  Interventions: Drug: Delgocitinib cream vehicle

INTERVENTIONS:
Drug: Delgocitinib cream — Cream for topical application
  Other Names: LEO 124249 cream
  Arms: Delgocitinib cream 1 mg/g; Delgocitinib cream 20 mg/g; Delgocitinib cream 3 mg/g; Delgocitinib cream 8 mg/g
Drug: Delgocitinib cream vehicle — The cream vehicle is similar to the delgocitinib cream except that it does not contain any active ingredient.
  Other Names: LEO 124249 cream vehicle
  Arms: Delgocitinib cream vehicle

SUMMARY:
This is a double-blind, multi-centre, randomised, 5-arm, vehicle-controlled, parallel-group trial. The trial is designed to establish a dose-response signal and investigate the efficacy and safety of delgocitinib cream in the treatment of adult subjects with mild to severe atopic dermatitis (AD).

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 years and above.
* Diagnosis of AD as defined by the Hanifin and Rajka 1980 criteria for AD.
* History of AD for ≥1 year.
* AD involvement of 5-50% treatable body surface area at screening and at baseline (excluding scalp).
* Disease severity graded as mild to severe according to vIGA-AD (i.e. vIGA-AD ≥2) at screening and baseline.

Key Exclusion Criteria:

* AD lesion(s) on scalp at screening and/or baseline.
* Active dermatologic conditions that may confound the diagnosis of AD or would interfere with assessment of treatment, such as scabies, cutaneous lymphoma, rosacea, urticaria, or psoriasis.
* Known active allergic or irritant contact dermatitis that is likely to interfere with the assessment of severity of AD.
* Use of tanning beds or phototherapy within 4 weeks prior to baseline.
* Systemic treatment with immunosuppressive/modulating drugs or corticosteroids within 4 weeks prior to baseline or 3 or more bleach baths any week within 4 weeks prior to baseline.
* Treatment with topical corticosteroids, topical calcineurin inhibitors, topical phosphodiesterase-4 inhibitors, or oral antibiotics within 2 weeks prior to baseline.
* Change in systemic antihistamine therapy within 2 weeks prior to baseline i.e. the subjects must not start antihistamine treatment or change the current dosage regime within 2 weeks prior to baseline.
* Receipt of live attenuated vaccines within 4 weeks prior to baseline.
* Treatment with any marketed or investigational biologic agents within 6 months or 5 half-lives prior to baseline, or until cell counts return to normal, whichever is longer.
* History of any active skin infection within 1 week prior to baseline.
* Clinically significant infection (systemic infection or serious skin infection requiring parenteral treatment) within 4 weeks prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (28):
- United States (10):
  - Leo Pharma Investigational Site, Birmingham, Alabama
  - Leo Pharma Investigational Site, Encino, California
  - Leo Pharma Investigational Site, Los Angeles, California
  - Leo Pharma Investigational Site, Rolling Hills Estates, California
  - Leo Pharma Investigational Site, Santa Ana, California
  - Leo Pharma Investigational Site, Chicago, Illinois
  - Leo Pharma Investigational Site, Detroit, Michigan
  - Leo Pharma Investigational Site, New York, New York
  - Leo Pharma Investigational Site, High Point, North Carolina
  - Leo Pharma Investigational Site, Philadelphia, Pennsylvania
- Australia (7):
  - Leo Pharma Investigational Site, Carlton
  - Leo Pharma Investigational Site, Darlinghurst
  - Leo Pharma Investigational Site, East Melbourne
  - Leo Pharma Investigational Site, Hectorville
  - Leo Pharma Investigational Site 1, Kogarah
  - Leo Pharma Investigational Site, Kogarah
  - Leo Pharma Investigational Site, Woolloongabba
- Canada (11):
  - Leo Pharma Investigational Site, Calgary, Alberta
  - Leo Pharma Investigational Site, Edmonton, Alberta
  - Leo Pharma Investigational Site, Surrey, British Columbia
  - Leo Pharma Investigational Site, Winnipeg, Manitoba
  - Leo Pharma Investigational Site, Fredericton, New Brunswick
  - Leo Pharma Investigational Site, Mississauga, Ontaria
  - Leo Pharma Investigational Site, Barrie, Ontario
  - Leo Pharma Investigational Site, Markham, Ontario
  - Leo Pharma Investigational Site, Peterborough, Ontario
  - Leo Pharma Investigational Site, Richmond Hill, Ontario
  - Leo Pharma Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 251 participants from 31 sites in 3 countries (U.S., Canada and Australia) were randomised in this trial. The first participant was screened on 29-Nov-2018 and the last participant completed the trial on 19-May-2020.
Pre-assignment Details: 326 participants were screened for this trial. Of these, 75 participants (23.0%) were screening failures. The main reason for screening failure was failure to meet eligibility criteria (18.4%).
Period: Overall Study
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Started (Number of subjects randomized) | 49 | 50 | 50 | 52 | 50
Completed | 38 | 44 | 44 | 46 | 36
Not Completed | 11 | 6 | 6 | 6 | 14
Not completed — Lack of Efficacy | 2 | 1 | 2 | 0 | 2
Not completed — Adverse Event | 2 | 2 | 1 | 0 | 6
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 4 | 4
Not completed — Lost to Follow-up | 3 | 1 | 2 | 2 | 1
Not completed — Personal reasons | 0 | 0 | 1 | 0 | 1
Not completed — COVID-19 situation | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of subjects randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle | Total
Number analyzed (Participants) | 49 | 50 | 50 | 52 | 50 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (16.1) | 38.5 (16.6) | 42.0 (17.4) | 37.4 (14.7) | 41.3 (19.6) | 40.5 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 32 | 37 | 36 | 172
  Male | 15 | 17 | 18 | 15 | 14 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 8 | 1 | 25
  Not Hispanic or Latino | 44 | 44 | 45 | 44 | 49 | 226
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 28 | 23 | 28 | 26 | 132
  Black or African American | 3 | 11 | 5 | 4 | 8 | 31
  Asian | 12 | 9 | 19 | 15 | 14 | 69
  Native Hawaiian or other Pacific islander | 0 | 0 | 0 | 0 | 1 | 1
  American Indian or Alaska native | 0 | 0 | 0 | 1 | 0 | 1
  Other | 7 | 2 | 3 | 4 | 1 | 17
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 9 | 19 | 15 | 14 | 72
  United States | 23 | 29 | 19 | 24 | 25 | 120
  Australia | 11 | 12 | 12 | 13 | 11 | 59
Baseline EASI score [Mean (Standard Deviation); unit: units on a scale] — EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe or more extensive condition.
  units on a scale | 9.3 (5.2) | 10.9 (9.1) | 8.6 (4.6) | 9.9 (6.9) | 11.2 (7.3) | 10.0 (6.8)
Baseline vIGA-AD score [Count of Participants; unit: Participants] — vIGA-AD is an instrument used in clinical trials to assess the subject's global disease severity and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    0 - Clear | 0 | 0 | 0 | 0 | 0 | 0
    1 - Almost clear | 0 | 0 | 0 | 0 | 0 | 0
    2 - Mild | 18 | 18 | 18 | 19 | 17 | 90
    3 - Moderate | 27 | 28 | 28 | 28 | 29 | 140
    4 - Severe | 4 | 4 | 4 | 5 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 0) to Week 8 in Eczema Area and Severity Index (EASI) Score.
Description: EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe or more extensive condition.
  The multiple comparison procedure - modelling (MCP-Mod) approach was used to guide dose selection. Mixed Model for Repeated Measurements (MMRM) analysis was used to determine the difference in the continuous endpoint between the active delgocitinib doses and delgocitinib cream vehicle.
Time Frame: Week 0 to Week 8
Population: FAS (defined as all randomized subjects exposed to investigational medicinal product)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 49 | 50 | 50 | 51 | 50
score on a scale | -5.0 (0.7) | -4.9 (0.7) | -5.8 (0.7) | -7.6 (0.7) | -1.9 (0.8)
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream 3 mg/g vs Delgocitinib Cream 8 mg/g vs Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; The primary endpoint was evaluated by determining if there was a dose-response relationship between the change from baseline to Week 8 in EASI score and the dose administered using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed and multiple comparison techniques were used to choose the model(s) likely to present the true underlying dose-response curve; Test type: Superiority; p < 0.0001, Multiple contrast test — P-values were adjusted for multiple comparisons. Models with adjusted p-value of <0.025 were stat. sign. diff. from a flat dose-response model. Model selected: Sigmoid Emax model
Statistical Analysis 2: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; Least square (LS) means were calculated using a mixed model response model (MMRM) on post-baseline responses up to Week 8 with an unstructured covariance matrix, Kenward-Roger approximation to estimate denominator degrees of freedom and the mean modelled as follows: Change from baseline in EASI = treatment x visit + baseline EASI x visit + region + baseline vIGA-AD. The primary comparison between each active delgocitinib dose and delgocitinib cream vehicle was at Week 8; Test type: Superiority; p < 0.01, Mixed Models Analysis — The stat. test was not controlled for multiplicity. Data at visits following premature discont. of IMP or initiation of rescue med. were excluded from the analysis. Likewise for missing data due to COVID-19 pandemic; Mean Difference (Net) = -3.1, 95% CI 2-sided [-5.0 to -1.3]
Statistical Analysis 3: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -3.0, 95% CI 2-sided [-4.8 to -1.2]
Statistical Analysis 4: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = -4.0, 95% CI 2-sided [-5.8 to -2.1]
Statistical Analysis 5: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Median Difference (Net) = -5.7, 95% CI 2-sided [-7.5 to -3.9]

2. Secondary Outcome: Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) Score of 0 (Clear) or 1 (Almost Clear) With ≥2-step Improvement (vIGA-AD TS) From Baseline to Week 8.
Description: vIGA-AD is an instrument used in clinical trials to assess the subject's global disease severity and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  The multiple comparison procedure - modelling (MCP-Mod) approach was used to guide dose-selection. Cochran-Mantel-Haenszel analysis was used to determine the difference in response rates between the active delgocitinib cream doses and the delgocitinib cream vehicle.
Time Frame: Week 0 to Week 8
Population: FAS (defined as all randomized subjects exposed to investigational medicinal product).
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 49 | 48 | 50 | 50 | 48
Participants | 9 | 14 | 15 | 24 | 5
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream 3 mg/g vs Delgocitinib Cream 8 mg/g vs Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; This endpoint was evaluated by determining if there was a dose-response relationship between the vIGA-AD response rate at Week 8 and the dose administered using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed and multiple comparison techniques were used to choose the model(s) most likely to represent the true underlying dose-response; Test type: Superiority; p < 0.0001, Multiple contrast test — Data collected after premature discont. of IMP due to COVID-19 were set to missing Week 8. Data collected after premature discont. of IMP due to reasons unrelated to COVID-19 or due to initiation of rescue med. were imputed as non-responders; P-values adj. for multiple comparisons. Models with adj. p-value <0.025 were stat. sign. diff. from a flat dose-response model. Model: Linear model
Statistical Analysis 2: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; The difference in response rates between the active delgocitinib cream doses and delgocitinib cream vehicle was analysed separately for each of the active dose groups using the Cochran-Mantel-Haenszel test stratified by region and disease severity (baseline vIGA-AD score). The null hypothesis of no difference in response rates between the delgocitinib cream active doses and delgocitinib cream vehicle was tested against the 2-sided alternative test that there is a difference; Test type: Superiority; p > 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 8.2, 95% CI 2-sided [-5.6 to 21.9]
Statistical Analysis 3: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 19.3, 95% CI 2-sided [3.9 to 34.6]
Statistical Analysis 4: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 20.3, 95% CI 2-sided [5.4 to 35.2]
Statistical Analysis 5: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 38.3, 95% CI 2-sided [22.3 to 54.3]

3. Secondary Outcome: EASI75 at Week 8
Description: EASI75 is defined as at least 75% reduction in EASI from baseline.
Time Frame: Week 0 to Week 8
Population: FAS (defined as all randomized subjects exposed to investigational medicinal product).
Measure: Count of Participants; unit: Participants
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 49 | 48 | 50 | 50 | 48
Participants | 20 | 21 | 28 | 33 | 10
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream 3 mg/g vs Delgocitinib Cream 8 mg/g vs Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; This endpoint was evaluated by determining if there was a dose-response relationship between EASI75 at Week 8 and the dose administered using the Multiple Comparison Procedure - Modelling (MCP-Mod) methodology. Several candidate parametric models were assumed and multiple comparison techniques were used to choose the model(s) most likely to represent the true underlying dose-response; Test type: Superiority; p < 0.0001, Multiple contrast test — [p-value comment as in outcome 2, analysis 1]; P-values were adj. for multiple comparisons. Models with adj. p-value <0.025 were stat. sign. diff. from a flat dose-response model. Model:Emax model
Statistical Analysis 2: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 19.7, 95% CI 2-sided [1.8 to 37.6]
Statistical Analysis 3: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 23.5, 95% CI 2-sided [5.8 to 41.2]
Statistical Analysis 4: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 35.3, 95% CI 2-sided [17.5 to 53.2]
Statistical Analysis 5: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Difference (RD) = 45.4, 95% CI 2-sided [28.1 to 62.8]

4. Secondary Outcome: Time to vIGA-AD TS
Description: The time to vIGA-AD TS response is defined as the time from baseline to first assessment of a vIGA-AD score of 0 (Clear) or 1 (Almost Clear) with ≥2-step improvement
Time Frame: Week 0 to Week 8
Population: FAS (defined as all randomized subjects exposed to investigational medicinal product)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
Number analyzed (Participants) | 49 | 50 | 50 | 51 | 50
Days | 64 [42 to 64] | NA [42 to NA] — The median time to achieve success in vIGA-AD was not estimable as fewer participants (less than 50%) reached success in vIGA-AD. | 64 [28 to 64] | 44 [26 to NA] — The 75% quartile to achieve success in vIGA-AD was not estimable as fewer participants (less than 75%) reached success in vIGA-AD. | NA [56 to NA] — The median time to achieve success in vIGA-AD was not estimable as fewer participants (less than 50%) reached success in vIGA-AD.
Statistical Analysis 1: Comparison: Delgocitinib Cream 1 mg/g vs Delgocitinib Cream Vehicle; Time to vIGA-AD TS was def. as time from date of first IMP applic. to first assess. of vIGA-AD TS. Subjects without baseline observation were censored at date of first IMP applic. Subjects with baseline observation not achieving vIGA-AD TS during treatment period were censored at date of last visit with a valid post-baseline assess. on or prior to date of discont. of IMP or initiation of rescue med, whichever occurred first. Subjects affected by COVID-19 pandemic were handled in the same manner; Test type: Other — Treatment groups were compared using a 2-sided log-rank test stratified by region and baseline vIGA-AD score. An event was defined as the first time achieving vIGA-AD; p > 0.05, Log Rank — The statistical test was not controlled for multiplicity
Statistical Analysis 2: Comparison: Delgocitinib Cream 3 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p > 0.05, Log Rank — vIGA-AD was reached in less than 50% of participants, therefore the median time was not estimable. The statistical test was not controlled for multiplicity
Statistical Analysis 3: Comparison: Delgocitinib Cream 8 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p > 0.05, Log Rank — The statistical test was not controlled for multiplicity
Statistical Analysis 4: Comparison: Delgocitinib Cream 20 mg/g vs Delgocitinib Cream Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p < 0.001, Log Rank — The statistical test was not controlled for multiplicity

ADVERSE EVENTS:
Time Frame: 10 weeks (from first application of IMP up until the last visit (safety follow-up visit)).
Description: Adverse events reported for all randomized subjects exposed to investigational medicinal product
Arm/Group | Delgocitinib Cream 1 mg/g | Delgocitinib Cream 3 mg/g | Delgocitinib Cream 8 mg/g | Delgocitinib Cream 20 mg/g | Delgocitinib Cream Vehicle
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/50 | 0/50 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/50 | 0/50 | 0/51 | 1/50
Other Adverse Events (participants affected / at risk) | 12/49 | 11/50 | 8/50 | 12/51 | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream 1 mg/g (N=49) | Delgocitinib Cream 3 mg/g (N=50) | Delgocitinib Cream 8 mg/g (N=50) | Delgocitinib Cream 20 mg/g (N=51) | Delgocitinib Cream Vehicle (N=50)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delgocitinib Cream 1 mg/g (N=49) | Delgocitinib Cream 3 mg/g (N=50) | Delgocitinib Cream 8 mg/g (N=50) | Delgocitinib Cream 20 mg/g (N=51) | Delgocitinib Cream Vehicle (N=50)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 3 (4) | 6 (6) | 6 (8) | 4 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 3 (4)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma A/S seeks publication of all clinical trials in peer-reviewed journals within 18 months after completion or termination of the clinical trial, regardless of whether the findings are positive or negative. After such a publication is made public, or if no publication is submitted by LEO Pharma A/S within these 18 months, the investigator has the right to publish the results from the clinical trial generated by him/herself.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03725722/Prot_SAP_000.pdf